CLINICAL TRIAL: NCT03719729
Title: A Phase II Study of Rifaximin (Xifaxan) for Patients With Sickle Cell Disease (SCD)
Brief Title: Rifaximin to Modify the Disease Course in Sickle Cell Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-12648
Record Dates: First submitted 2018-09-04; First posted 2018-10-25 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-08

CONDITIONS: Sickle Cell Disease; Antibiotics
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Each subject will receive rifaximin 550 mg twice a day for up to one year.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Administer daily rifaximin to modify intestinal microbiome to alter the course of the disease.
  Other Names: Xifaxan

SUMMARY:
In this single-arm, one-stage Phase II study, the investigators hypothesize that gut decontamination with rifaximin will reduce the frequency of hospital admission due to painful crisis in patients with SCD. The study will accrue 20 SCD patients who had at least two hospital admissions in the previous 12 months. These patients will receive rifaximin 550 mg twice a day for a total of 12 months. This following clinical parameters will be measured: 1. Changes in the annual rate of hospital admissions due to painful crisis; 2. Changes in the annual rate of days hospitalized; 3. Annual rates of uncomplicated crises; 4. Annual rate of acute chest syndrome; 5. Changes in the quality of life; and 6). Toxicities. The following laboratory parameters will be measured: 1. Changes in the number of circulating activated neutrophils; 2. Changes in the intestinal microbiome diversity; 3. Changes in the urinary 3-indoxyl sulfate levels; 4. Changes in the serum biomarkers of intestinal permeability (lipopolysaccharides; zonulin, citrulline, and fatty acid binding proteins).

DETAILED DESCRIPTION:
In this single-arm Phase II study, the investigators will accrue 20 SCD patients who had at least two hospital admissions in the previous 12 months to receive rifaximin 550 mg twice a day for a total of 12 months. The investigators will measure changes in the annual rate of hospital admissions due to vaso-occlusive crisis and the annual rate of hospital days. The investigators will also determine the annual rates of uncomplicated crises and acute chest syndrome. Quality of life due to the disease and to treatment will be determined using a questionnaire. This study will be complemented with exploratory laboratory studies to determine changes in the number of circulating activated neutrophils, intestinal microbiome diversity, urinary 3-indoxyl sulfate levels and serum biomarkers of intestinal permeability (lipopolysaccharides; zonulin, citrulline, and fatty acid binding proteins).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HbSS, HbSC, or HbS beta thal.
2. Age 18-70 years.
3. More than two hospital admissions for painful VOC in the prior 12 months, whether on any anti-sickling agents (e.g. hydroxyurea, L-glutamine, or transfusion therapy) or not. These agents may be continued during the study period. However, subjects are not allowed to be started on any of these agents during the study period.
4. Ability to comprehend and sign an informed consent. -

Exclusion Criteria:

1. Pregnant or lactating. For female subjects of child-bearing potential, the subject must agree to avoid pregnancy during the rifaximin study period and to practice a recognized form of birth control during this period (e.g. barrier, birth control pills, abstinence).
2. Life expectancy of < 12 months.
3. History of allergy to rifaximin.
4. Patients with newly developed abnormal vital signs or abnormal physical examination (outside the signs that are expected in patients with SCD).
5. Patients in active VOC.
6. Patients with a baseline prothrombin time International Normalized ratio (INR) >2.0.
7. Patients who receive any blood products within three weeks of the screening visit.
8. Patients with uncontrolled liver disease or renal insufficiency, colitis, or inflammatory bowel disease.
9. Patients with HIV, or other concomitant immunodeficiency.
10. Patients on penicillin prophylaxis or antibiotics for treatment of infection.
11. Patients with significant medical condition that require hospitalization (other than sickle cell VOC) within two months of the screening visit.
12. Patients currently taking or has been treated with an investigational drug within 30 days of the screening visit.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-02-22 (Estimated); Study Completion 2020-07-22 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile | 24 months
  Incidence of nausea, vomiting, diarrhea, abdominal discomfort, worsening anemia.

SECONDARY OUTCOMES:
Changes in the annual rate of hospital admission for painful crisis | 12 months
  Changes in the frequency of hospitalization for painful crisis
Changes in the annual days of hospitalization for painful crisis | 12 months
  Changes in the total number of days in hospital due to painful crisis
Changes in the annual number of units of blood transfusion | 12 months
  Changes in the number of units of blood transfused
Changes in the quality of life as measured by the FANLTC questionnaire | 24 months
  Changes in the quality of life due to treatment with rifaximin

CONTACTS AND LOCATIONS:
Locations (1):
- Westchester Medical Cancer Cancer Institute, Valhalla, New York, United States